CLINICAL TRIAL: NCT01069822
Title: A Phase I Open-label, Fixed Sequence Study to Determine the Effect of Multiple Intravenous Doses of AZD6765 on the Pharmacokinetics of Oral Midazolam (CYP3A4 Substrate) in Healthy Subjects
Brief Title: A Study in Healthy Volunteers to Assess Effect of AZD6765 on Midazolam Blood Levels
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: D6702C00008
Record Dates: First submitted 2010-02-15; First posted 2010-02-17 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
Keywords: Midazolam; Pharmacokinetics
MeSH Terms: interventions — AZD6765; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): midazolam + AZD6765 IV solution
  Interventions: Drug: AZD6765; Drug: midazolam
- 2 (Active Comparator)
  Interventions: Drug: midazolam

INTERVENTIONS:
Drug: AZD6765 — IV solution
  Arms: 1
Drug: midazolam

SUMMARY:
The main purpose of this study is to evaluate the effect repeated doses of AZD6765 (a drug being developed for the treatment of patients with severe major depressive disorder) has on the PK (pharmacokinetic) profile of Midazolam. (The PK profile is how the drug leaves your body and acts in the body.)

ELIGIBILITY:
Inclusion Criteria:

* BMI between 19-30

Exclusion Criteria:

* Significant result for C-SSRS at screening or baseline
* Single arm preference for IV procedures

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2010-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters to be calculated from midazolam and AZD6765 plasma concentrations | on Day -1 and Day 6

SECONDARY OUTCOMES:
Safety variables (adverse events, vital signs, physical and neurological examinations, clinical laboratory assessments, 12-lead ECG, C-SSRS, CADSS, and VAS scales) | will be collected from the time of informed consent (Visit 1) until completion of the follow-up visit.
Optional Genetic sampling | at admission Day -2
Exploratory - renal biomarkers in urine | At admission Day -2 until follow up visit

CONTACTS AND LOCATIONS:
Overall Officials: Willie Earley, MD, Study Director — AstraZeneca; Brendan Smyth, MD, Ph.D, Study Director — AstraZeneca; Phil Leese, MD, Principal Investigator — Quintiles, Inc.
Locations (1):
- Research Site, Overland Park, Kansas, United States

REFERENCES:
- See also: D6702C00008 Clinical Study Report Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=572&filename=D6702C00008_Clinical_Study_Report_Synopsis.pdf